CLINICAL TRIAL: NCT01299857
Title: EVALUATION CLINIQUE ET BIOLOGIQUE A LONG TERME DES PATIENTS ATTEINTS DE FORMES SEVERES DE PEMPHIGUS TRAITES PAR LE RITUXIMAB
Brief Title: Long-term Clinical and Biological Evaluation of Patients With Severe Forms of Pemphigus Treated by Rituximab
Acronym: Suiviritux
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 2009/141/HP
Record Dates: First submitted 2011-02-17; First posted 2011-02-18 (Estimated); Last update posted 2012-09-13 (Estimated); Status verified 2012-09

CONDITIONS: Pemphigus
Keywords: pemphigus; Mabthéra (R); B lymphocytes; desmogleines
MeSH Terms: conditions — Pemphigus | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Rituximab — 375mg/m2
  Other Names: Mabthéra

SUMMARY:
The purpose of this study is to study the midterm clinical evaluation, biological parameters and immune reconstitution after Rituximab treatment for Pemphigus.

ELIGIBILITY:
Inclusion Criteria:

* age>18
* consentment
* patient treated with Rituximab and included in clinical trial n°2002/020/HP - NCT00213512 "Treatment of Patients Presenting Pemphigus With Anti CD20 (Mabthera)".

Exclusion Criteria:

* age < 18
* no consentment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2011-06; Primary Completion 2011-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Rate of relapse after 5 years of treatment | five years
  Primary outcome measure is the evaluation of Rate of relapse after 5 years of treatment by rituximab for patient with pemphigus. The relapse is defined by the reappearance of mucous or cutaneous érosives lésions proved by histology and by direct immunofluorescence

CONTACTS AND LOCATIONS:
Overall Officials: Damien PICARD, Doctor, Principal Investigator — dermatological department
Locations (1):
- UH-Rouen, Rouen, Seine maritime,, France